CLINICAL TRIAL: NCT02781909
Title: Pilot Study to Estimate the Potential Efficacy and Safety of Using Adjunctive Ibuprofen for the Treatment of XDR Tuberculosis
Brief Title: Potential Efficacy and Safety of Using Adjunctive Ibuprofen for XDR-TB Tuberculosis
Acronym: NSAIDS-XDRTB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSAIDS4TB_01
Record Dates: First submitted 2016-05-02; First posted 2016-05-25 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Tuberculosis
Keywords: NSAIDS; tuberculosis treatment; anti-inflammatories; Host-directed therapies; TB
MeSH Terms: conditions — Tuberculosis | interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: Standard of Care TB treatment (Active Comparator): Individuals with confirmed pulmonary XDR-TB and receiving Standard of Care TB treatment according to national and WHO guidelines; n=12
  Interventions: Drug: Standard of Care TB treatment
- Ibuprofen-treated (Experimental): Individuals with confirmed pulmonary XDR-TB and receiving Standard of Care TB treatment according to national and WHO guidelines plus ibuprofen (400mg/day/2 months); n=12
  Interventions: Drug: Ibuprofen; Drug: Standard of Care TB treatment

INTERVENTIONS:
Drug: Ibuprofen — Non-Steroid Anti-Inflammatory drug to be administered as adjunctive therapy
  Other Names: NSAID
  Arms: Ibuprofen-treated
Drug: Standard of Care TB treatment — Standard of Care (SoC) TB Treatment will be optimized and drugs selected according to the National and WHO Guidelines, sensitivity profile and as per routine.
  Other Names: anti-TB treatment

SUMMARY:
Novel approaches to improve TB treatment outcomes (to reduce morbidity, mortality, and the duration of TB treatment) and to treat XDR-TB cases are urgently required. Host-Directed therapies (especially repurposed drugs such as Non-Steroid AntiInflammatory Drugs NSAIDS) could be useful in this context, and therefore the appropriateness and potential effect of this approach needs to be evaluated in humans. Investigators do propose a prospective, randomized, pilot study to estimate the potential efficacy and safety of using adjunctive ibuprofen for the treatment of XDR tuberculosis.

DETAILED DESCRIPTION:
There are a need for novel approaches to improve TB treatment outcomes (to reduce morbidity, mortality, and the duration of TB treatment) and to treat XDR-TB cases. Host-Directed therapies (especially repurposed drugs such as Non-Steroid AntiInflammatory Drugs NSAIDS) could be useful in this context, and therefore the appropriateness and potential effect of this approach needs to be evaluated in humans. Investigators do propose a prospective, randomized, pilot clinical trial to evaluate the potential efficacy and safety of using adjunctive ibuprofen during two months for the treatment of XDR tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males aged ≥ 16
2. The patient must provide written informed consent
3. Females of childbearing potential (including females less than 2 years post- menopausal) must have a negative pregnancy test at enrolment and must agree to use highly effective methods of birth control
4. M.tuberculosis (Mtb) detected by culture with available drug susceptibility results for current isolate
5. XDR- TB confirmed by drug susceptibility testing (DST)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Inability to provide written informed consent
2. First line drug treatment susceptible Mtb strain
3. Prior Treatment of either >3 days of TB treatment prior to randomization
4. Pregnancy/Breastfeeding at inclusion
5. Any of the following laboratory parameters: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN); total bilirubin > 2 x ULN; estimated glomerular filtration rate (eGFR) <60ml/hr; Neutrophil count ≤ 500 neutrophils / mm3; Platelet count < 50,000 cells / mm3
6. Receiving or anticipated to receive a daily dose of ≥ 10 mg of systemic prednisone or equivalent within the period starting 14 days prior to enrolment, or > 5 doses per week of any NSAID for ≥2 weeks in the month prior to randomization.
7. History of sensitivity or allergy to ibuprofen.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of pilot study participants with microbiological efficacy-related events that are related to treatment. | 6 months
  Number of pilot study participants with negative sputum culture at M2 and M6 following inclusion
Number of pilot study participants with radiological efficacy-related events that are related to treatment. | 6 months: at baseline, at month 3 and month 6
  Changes detected by X-ray during follow-up up to month 6
Number of pilot study participants with clinical efficacy-related events that are related to treatment. | 6 months
  Final treatment outcomes according to the WHO definitions including all time in follow-up to M6 on TB treatment
Microbiological efficacy-related events: Time to stable culture conversion up to M6 | 6 months
  Time to stable culture conversion up to M6: (≥ two consecutive cultures negative for M. tuberculosis) including all time in follow-up to month six on TB treatment. Differences between the two groups

SECONDARY OUTCOMES:
Number of pilot study participants with Safety-related events. | 6 months
  Outcome measurements: incidence of safety-related events during the whole study period: clinical worsening of the disease, no sputum conversion (if AFS-), any worsening concerning vital parameters and routine blood work.
Proportion of pilot study participants showing differences in Health Quality of Life (HQoL). | 2 and 6 months
  Outcome measurements: HQoL measures at M2 and M6 relative to baseline.
Proportion of pilot study participants showing differences in Immune Responses at M2 and M6 relative to baseline. | 2 and 6 months
  Outcome measurements: changes detected in immune responses at M2 and M6.

CONTACTS AND LOCATIONS:
Overall Officials: Cris Vilaplana, MD, PhD, Principal Investigator — Fundació Institut Germans Trias i Pujol
Locations (2):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Perinatal HIV Unit (PHRU), Soweto, South Africa

REFERENCES:
- See also: Experimental Tuberculosis Unit of the Germans Trias i Pujol website (PI's affiliation) — https://unitatdetuberculosiexperimental.wordpress.com/
- See also: Host-Directed Therapies Network website — http://www.unza-uclms.org/hdt-net